CLINICAL TRIAL: NCT05318482
Title: Effects of Physical Activity of an In-hospital Motivational Program in Cardio-respiratory Patients: a Randomized Control Trial
Brief Title: Motivational Program on Physical Activity in Cardio-respiratory Patients: an RCT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CE 2608
Record Dates: First submitted 2022-03-30; First posted 2022-04-08 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Cardiorespiratory Failure
Keywords: Rehabilitation; behaviour; COPD; heart failure; tracing
MeSH Terms: conditions — Behavior; Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Cardio-respiratory patients (COPD and CHF), with similar comorbidity, needing rehabilitation, will be consecutively enrolled at Istituti Clinici Scientifici Maugeri.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational group (Experimental): The patients of this group will be equipped with an electronic wristwatch and will be monitored every day by the physiotherapist (PT) through an application on their mobiles. The PT will follow these patients with a daily motivational session (15 minutes, modality 1 patient: 1 PT) and with an educational program about the definition, importance and benefits of physical activity.
  Interventions: Behavioral: Motivational group
- Control (Sham Comparator): The patients of this group will have an electronic wristwatch and will be advised by the PT only with generic recommendations of daily exercise during the hospitalization, besides the usual activities of the rehabilitation program.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Motivational group — In addition to the activities of the usual rehabilitation program, the PT will perform a daily motivational session of 15 minutes in a 1 patient: 1 physiotherapist modality. On that occasion, the patient will report the number of steps performed the previous day; the physiotherapist will check and promote the increase of 10% in the number of steps for the next day. If the patient fails to achieve the goal, the PT will analyze the reasons with the patient, in order to facilitate the achievement of the goal. The PT will advise on the time and place to perform physical activity and the patients will receive a diary to record his/her progress (number of steps and heart rate, Borg Fatigue and Borg Dyspnea before and after an exercise task). The PT will record all these evaluations on an excel database.
  Arms: Motivational group
Other: Control group — Besides the activities of the usual rehabilitation program, the patients of this group will be provided by the PT only with the generic recommendations of daily exercise during the in-hospital stay
  Other Names: Generic recommendations
  Arms: Control

SUMMARY:
According to actual scientific evidence, the interventions on the general population aiming at regular physical activity are one of the most efficient strategies for health improvement. Regardless of this evidence, there is a large part of the elderly population does not adhere to the recommendations of the international guidelines on daily physical activity.

This is even more evident in patients with chronic respiratory and cardiological disease because exercise exacerbates existing symptoms of breathlessness.

This study aims to evaluate the impact of an in-hospital motivational program dedicated to increasing physical activity. With the data of an electronic wristwatch that keeps records of movement, the health professionals incentive an increase in physical activity leading to long term behavioural changes (evaluated by the number of steps per day) in hospitalized patients with COPD and HF, which already perform a standard rehabilitation program (14 sessions).

DETAILED DESCRIPTION:
There are studies in the literature that have reported, in comparison with healthy subjects, a lower level of physical activity in COPD patients; other studies associate less physical activity with increased risk of hospitalization and mortality, which is even more evident considering patients with chronic respiratory diseases. In the same way, patients with Heart Failure (HF) reduce their activity and exercise capacity increasing hospitalization and mortality.

With more fatigue and dyspnoea, a vicious circle is created, with a consequent further reduction of levels of physical activity and worsening of symptoms.

Therefore, it is necessary to provide augmented physical activity in rehabilitation hospital environments.

Rehabilitation is a way to encourage and support patients to achieve their best physical condition. At present, COPD and HF patients admitted in rehabilitative cardio-respiratory wards dedicate a limited amount of time to physical activity, when referred to the entire day of hospitalization, whereas the rest of their time is spent in a sedentary condition. Thus, it is difficult to imagine that an actual change in the patients' lifestyle can be obtained by such a cardio-respiratory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* >18 years, both of genders;
* Scheduled time of hospitalization of at least 14-16 days;
* Ability to walk by themselves, with safety (SPPB >10);
* Hospital admission with a diagnosis of COPD (GOLD III-IV, B-D), with or without respiratory failure, or HF (NYHA II-III), sufficiently stabilized with a specific pharmacological therapy
* Possession of a smartphone and ability to use the app for health tracking.

Exclusion Criteria:

* Significant symptoms of the primary disorder, not properly stabilized;
* Hemodynamic and clinic instability;
* Musculoskeletal issues or other types (neurological, orthopedical…), which involve an important limitation in physical exercise performance;
* Medical comorbidities with a life expectancy shorter than one year;
* Clinical signs of cognitive impairment (MMSE < 25).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Delta change in number of steps per day | Day 0 and day 17
  To evaluate the impact of a motivational program, by an electronic wristwatch for health tracking dedicated to improving physical activity, on behavioural changes (number of steps per day) in hospitalized patients with COPD and HF, which already have performed a standard rehabilitation program.

SECONDARY OUTCOMES:
Delta change in PASE Questionnaire | Day 0 and day 17
  The Physical Activity Scale for the Elderly (PASE) is an easily administered and scored instrument that measures the level of physical activity in individuals aged 65 years and older. It is divided into two main sections, one for the activities performed in the spare time, and one for household activities. The total score is obtained by multiplying the time amount spent on each free-time activity (hours/day/week) or household activity (yes/no) by certain values derived empirically for each of them; the sum of all activities correlates with the physical activity level.
Delta change in 6 MWT | Day 0 and day 17
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  This assessment will include also the Borg Scale for Dyspnoea and Fatigue. They both have a minimum score, 0, and a maximum score, 10. Higher scores indicate greater symptom severity (either for dyspnoea or for fatigue).
Delta change in SPPB Scale | Day 0 and day 17
  The SPPB Scale evaluates the level of safety in motor ability. It is divided into three items, each ranging from 0 to 4. The first item is balance (the score is assigned according to the difficulty level in keeping balance), the second is walking (the score reflects the amount of time taken to walk a distance of 4 meters), and the third is the 1-Minute-Sit-To-Stand-Test (the score is determined by the number of lifts from sitting to standing, performed within the first 5 seconds in one minute. The sum of the scores for each item may vary from 0, which indicates the complete motor inability, to a maximum of 12, which indicates a total motor autonomy.
Delta change in EMI-2 questionnaire | Day 0 and day 17
  The EMI (Markland and Hardy, 1993) was developed as a means of assessing participation motives in order to examine such issues as the influence of motives on exercise participation, how such motives might influence the choice of activities undertaken, how affective responses to exercise may be influenced by reasons for exercising and how involvement in physical activity might have a reciprocal influence on participation motives. In particular, the authors developed the instrument to examine questions concerning the functional significance of exercise motives from the perspective of Deci and Ryan's (1985) self-determination theory. It is presented as a list of 51 motivational sentences, each of them is assigned a score from 0 (totally false) to 5 (totally true). The sum of each score is the final result, ranging from a minimum of 0 (absence of motivation to do exercise) to a maximum of 255 (highest motivation to do exercise).
Delta change in SF-12 questionnaire | Day 0 and day 17
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 uses the same eight domains as the SF-36:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The PCS includes 6 questions concerning different issues. Two questions are about physical activit
Delta change in BDI questionnaire | Day 0 and day 17
  The Beck Depression Inventory (BDI) is a 21-item self-reporting questionnaire for evaluating the severity of depression in normal and psychiatric populations.
  Twenty-one items were consolidated from those observations and ranked 0-3 for severity. The questionnaire is administered by health professionals. The minimum score is 0 and the maximum score is 63. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No
Protocol submitted to technical and Scientific Committee and Ethical Committee

REFERENCES:
- [Background] Demeyer H, Louvaris Z, Frei A, Rabinovich RA, de Jong C, Gimeno-Santos E, Loeckx M, Buttery SC, Rubio N, Van der Molen T, Hopkinson NS, Vogiatzis I, Puhan MA, Garcia-Aymerich J, Polkey MI, Troosters T; Mr Papp PROactive study group and the PROactive consortium. Physical activity is increased by a 12-week semiautomated telecoaching programme in patients with COPD: a multicentre randomised controlled trial. Thorax. 2017 May;72(5):415-423. doi: 10.1136/thoraxjnl-2016-209026. Epub 2017 Jan 30. PMID 28137918